CLINICAL TRIAL: NCT07002086
Title: The Effects of Tourniquet Applied to the Lower Extremity During Total Knee Replacement Surgery on Hemodynamics, ETCO2, SpO2 and Blood Picture of Patients
Brief Title: Effects of Tourniquet Applied During Total Knee Replacement Surgery on Patient Hemodynamics and Blood Table
Status: Completed | Type: Observational
Sponsor: Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Fatma Acil,MD, Principal Investigator, Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital
Other Study IDs: 67926
Record Dates: First submitted 2025-05-23; First posted 2025-06-03 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Primary Gonarthrosis
MeSH Terms: interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Total knee replacement — * Is a surgical procedure to resurface a knee damaged by arthritis. Metal and plastic parts are used to cap the ends of the bones that form the knee joint, along with the kneecap.
  * In the surgical procedure of these surgeries, cement is used to fix the prosthesis.
  Other Names: knee arthroplasty; Knee replacement

SUMMARY:
This study was planned to investigate the physiopathology of bradycardia and hypotension that occur in some patients with total knee arthroplasty (TKA) between the ages of 65 and 90 years when the tourniquet, which is routinely used in patients with total knee arthroplasty (TKA), is opened at the end of the operation and to determine the physiopathology of these effects of the tourniquet and how these effects can be prevented.

DETAILED DESCRIPTION:
This study was planned to investigate the effects of lower extremity tourniquets routinely used in TDP surgeries on hemodynamics, SpO2, ETCO2 and blood tables in male and female patients aged 65-90 years. In the patients included in the study, measurements from the monitor will be recorded and preop and postop hemogram, complete biochemistry, coagulation arterial blood gases will be recorded from each patient's file and the values before and after the tourniquet will be compared. New randomized prospective studies will be proposed by determining the physiopathological changes (reperfusion syndrome) that occur after opening the tourniquet in patients and evaluating how these changes can be prevented

ELIGIBILITY:
Inclusion Criteria:

* ASA score: 1-3
* primary gonarthrosis

Exclusion Criteria:

* ASA score 4 and above
* The diagnosis of secondary gonarthrosis
* Concomitant rheumatological disorders
* Concomitant peripheral vascular disease
* Concomitant malignant disease
* Presence of organ failure
* Having active infection
* Use of immunosuppressive drugs
* Having addiction to cigarettes, alcohol or drugs
* Use of anticoagulation medicine
* Presence of metabolic disease
* Presence of renal disease
* Presence of familial hemophagocytic syndrome
* Being unwilling to participate the study

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients undergoing knee replacement surgery
Sampling Method: Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2025-06-04 (Actual); Primary Completion 2025-12-26 (Actual); Study Completion 2026-01-07 (Actual)

PRIMARY OUTCOMES:
Activated Partial Thromboplastin Time(APTT) | Time 1:Preoperative 24th hour, Time 2: Approximately 10-15 minutes after placing cement during surgery, Time 3: Approximately 10-15 minutes after opening the intraoperative leg tourniquet, Time 4: Postoperative 12th hour, Time 5: Postoperative 24th hour
  The activated partial thromboplastin time (APTT) is a screening test which isolates the 'intrinsic' and 'common' pathways of the in vitro coagulation cascade model. Coagulation factors and cofactors within each pathway operate in concert to generate a fibrin clot end-point, the time taken to form the clot being the APTT.
Prothrombin Time (PT) | Time 1:Preoperative 24th hour, Time 2: Approximately 10-15 minutes after placing cement during surgery, Time 3: Approximately 10-15 minutes after opening the intraoperative leg tourniquet, Time 4: Postoperative 12th hour, Time 5: Postoperative 24th hour
  Prothrombin Time (PT) : is an assay for evaluating the extrinsic pathway and common pathway of coagulation
International Normalised Ratio (INR) | Time 1:Preoperative 24th hour, Time 2: Approximately 10-15 minutes after placing cement during surgery, Time 3: Approximately 10-15 minutes after opening the intraoperative leg tourniquet, Time 4: Postoperative 12th hour, Time 5: Postoperative 24th hour
  Measured value used to monitor treatment with anticoagulants and to provide information on how quickly the blood clots. INR value of 1 = no anticoagulation; INR value of 2 = coagulation is prolonged 2-fold; INR value of 3 = coagulation is prolonged 3-fold.
D-DİMER | Time 1:Preoperative 24th hour, Time 2: Approximately 10-15 minutes after placing cement during surgery, Time 3: Approximately 10-15 minutes after opening the intraoperative leg tourniquet, Time 4: Postoperative 12th hour, Time 5: Postoperative 24th hour
  D-dimer (or D dimer) is a dimer that is a fibrin degradation product (FDP), a small protein fragment present in the blood after a blood clot is degraded by fibrinolysis.

SECONDARY OUTCOMES:
C reactive protein (CRP) | Time 1:Preoperative 24th hour, Time 2: Approximately 10-15 minutes after placing cement during surgery, Time 3: Approximately 10-15 minutes after opening the intraoperative leg tourniquet, Time 4: Postoperative 12th hour, Time 5: Postoperative 24th hour
  C-reactive protein (CRP) is an annular pentameric protein found in blood plasma, whose circulating concentrations rise in response to inflammation
Procalcitonin | Time 1:Preoperative 24th hour, Time 2: Approximately 10-15 minutes after placing cement during surgery, Time 3: Approximately 10-15 minutes after opening the intraoperative leg tourniquet, Time 4: Postoperative 12th hour, Time 5: Postoperative 24th hour
  It is considered a biomarker specific to bacterial infections.
Ferritin | Time 1:Preoperative 24th hour, Time 2: Approximately 10-15 minutes after placing cement during surgery, Time 3: Approximately 10-15 minutes after opening the intraoperative leg tourniquet, Time 4: Postoperative 12th hour, Time 5: Postoperative 24th hour
  Ferritin is an iron storage protein that also plays a role in numerous other conditions, including inflammatory, neurodegenerative and malignant diseases.
D-dimer | Time 1:Preoperative 24th hour, Time 2: Approximately 10-15 minutes after placing cement during surgery, Time 3: Approximately 10-15 minutes after opening the intraoperative leg tourniquet, Time 4: Postoperative 12th hour, Time 5: Postoperative 24th hour
  D-dimer is a byproduct of the blood clotting and breakdown process.
Fibrinogen | Time 1:Preoperative 24th hour, Time 2: Approximately 10-15 minutes after placing cement during surgery, Time 3: Approximately 10-15 minutes after opening the intraoperative leg tourniquet, Time 4: Postoperative 12th hour, Time 5: Postoperative 24th hour
  Is a soluble protein present in blood plasma, from which fibrin is produced by the action of the enzyme thrombin.
Lactat | Time 1:Preoperative 24th hour, Time 2: Approximately 10-15 minutes after placing cement during surgery, Time 3: Approximately 10-15 minutes after opening the intraoperative leg tourniquet, Time 4: Postoperative 12th hour, Time 5: Postoperative 24th hour
  Lactate is a bi-product constantly produced in the body during normal metabolism and exercise
Mean arterial pressure | Time 1:Preoperative 24th hour, Time 2: Approximately 10-15 minutes after placing cement during surgery, Time 3: Approximately 10-15 minutes after opening the intraoperative leg tourniquet, Time 4: Postoperative 12th hour, Time 5: Postoperative 24th hour
  Mean arterial pressure (MAP) is the average arterial pressure throughout one cardiac cycle, systole, and diastole.
  Expressed in mmHg
Heart rate | Time 1:Preoperative 24th hour, Time 2: Approximately 10-15 minutes after placing cement during surgery, Time 3: Approximately 10-15 minutes after opening the intraoperative leg tourniquet, Time 4: Postoperative 12th hour, Time 5: Postoperative 24th hour
  Heart rate is the frequency of the heartbeat measured by the number of contractions of the heart per minute
Neutrophil to Lymphocyte Ratio | Time 1:Preoperative 24th hour, Time 2: Approximately 10-15 minutes after placing cement during surgery, Time 3: Approximately 10-15 minutes after opening the intraoperative leg tourniquet, Time 4: Postoperative 12th hour, Time 5: Postoperative 24th hour
  The neutrophil-to-lymphocyte ratio (NLR), calculated as a simple ratio between the neutrophil and lymphocyte counts measured in peripheral blood, is a biomarker which conjugates two faces of the immune system: the innate immune response, mainly due to neutrophils, and adaptive immunity, supported by lymphocytes
Interleukin 1 | Time 1:Preoperative 24th hour, Time 2: Approximately 10-15 minutes after placing cement during surgery, Time 3: Approximately 10-15 minutes after opening the intraoperative leg tourniquet, Time 5: Postoperative 24th hour
  It is an inflammatory cytokine that has various physiological functions and pathological significance, playing an important role in health and disease.
Interleukin 6 | Time 1:Preoperative 24th hour, Time 2: Approximately 10-15 minutes after placing cement during surgery, Time 3: Approximately 10-15 minutes after opening the intraoperative leg tourniquet, Time 5: Postoperative 24th hour
  Is a potent anti-inflammatory cytokine that plays a crucial, and often essential, role in preventing inflammatory and autoimmune pathologies.
Interleukin 10 | Time 1:Preoperative 24th hour, Time 2: Approximately 10-15 minutes after placing cement during surgery, Time 3: Approximately 10-15 minutes after opening the intraoperative leg tourniquet, Time 5: Postoperative 24th hour
  Is a soluble mediator with pleiotropic effects on inflammation, immune response and hematopoiesis.
Tumor necrosis factor alfa (TNF alfa) | Time 1:Preoperative 24th hour, Time 2: Approximately 10-15 minutes after placing cement during surgery, Time 3: Approximately 10-15 minutes after opening the intraoperative leg tourniquet, Time 4: Postoperative 12th hour
  Is a cytokine that has pleiotropic effects on various cell types and has been identified as a major regulator of inflammatory responses and plays a role in the pathogenesis of some inflammatory and autoimmune diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Fatma Acil, M.D., Principal Investigator — Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital; Abdulkadir Yektaş, Prof. Dr., Study Director — Siirt University
Locations (1):
- Saglik Bilimleri Universitesi Gazi Yasargil Training and Research Hospital, Diyarbakır, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
* after de-identification; all individual participant data collected during the research and the primary and secondary outcomes of the study.
  * data can be shared immediately after publication, no end date set.
  * case-by-case basis at the discretion of Primary Sponsor
  * data can be access subject to approvals by Principal Investigator (e-mail: fatma.acil@saglik.gov.tr)